CLINICAL TRIAL: NCT05592132
Title: Use of Virtual Reality in Pain Management During Invasive Gestures in Pediatric Oncology: Randomized Controlled Trial
Brief Title: Use of Virtual Reality in Pain Management in Pediatric Oncology
Acronym: DOREVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022/CHU/11
Record Dates: First submitted 2022-06-30; First posted 2022-10-24 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Pediatric Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: intervention plus standard care versus standard care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized in this arm will have the virtual reality headset associated to the standard care
  Interventions: Other: Virtual reality headset
- Standard care (No Intervention): patients randomized in this arm will have standard care.

INTERVENTIONS:
Other: Virtual reality headset — Each patient in this treatment group will use a virtual reality headset during 3 procedures. During each procedure, the pain level will be assessed and compared with the assessed group.
  Arms: Intervention

SUMMARY:
DOREVI is a monocentric randomized controlled study that will evaluate the efficacy of virtual reality helmets for pain prevention during invasive care on 78 oncologic pediatric patients. Two groups of children (between 6 and 11 and between 12 and 18 years old) will be randomized to use helmet plus standard care or standard care alone during invasive procedures (central venous catheter puncture, lumbar puncture, or bone marrow aspiration). The pain intensity will be evaluated using a visual analogic scale during three invasive procedures, and results will be compared between the patients with or without virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* patient who tolerates the virtual reality headset
* patient followed in pediatric oncology
* patient with a diagnosis of benign tumor or cancer
* patient who needs to have painful medical procedure during their treatment
* patient whose parents have signed the informed consent
* patient affiliated with social security or equivalent

Exclusion Criteria:

* patient with visual or hearing impairement
* patient with epilepsy or other neurological disease
* patient with psychiatric disease

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Self pain evaluation | before blood sampling on catheter with implantable chamber
  Pain will be assessed by the analogic visual scale (minimal score = 0 (no pain) , maximal score = 10 (maximal pain))

CONTACTS AND LOCATIONS:
Overall Officials: Yves REGUERRE, Principal Investigator — CHU de La Réunion
Locations (1):
- CHU de La Réunion, Saint-Denis, Reunion